CLINICAL TRIAL: NCT02046473
Title: 3D Sonographic Measurement of Volumetric Flow in Transjugular Intrahepatic Porto-Systemic Shunts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Paula Novelli M.D., Principal Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00054436
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Portal Hypertension; Liver Disease
MeSH Terms: conditions — Hypertension, Portal; Liver Diseases | interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Volumetric Flow in TIPS (Other): Subjects who have TIPS (transjugular intrahepatic porto-systemic shunts) have measurements taken to determine if someone has increased blood pressure in the portal vein of the liver (portal hypertension). Subjects who have a TIPS receive clinical ultrasounds every 3 months to determine if the TIPS is working properly.
  Interventions: Procedure: Volumetric Flow in TIPS

INTERVENTIONS:
Procedure: Volumetric Flow in TIPS — Subjects who have a TIPS (transjugular intrahepatic portal-systemic shunt) for portal hypertension will undergo a clinical 3D ultrasound to determine if the TIPS is working properly. Additional ultrasounds will be obtained during the subject's clinically ordered ultrasound(s). These measurements will be taken by using a second ultrasound probe (plastic hand held device that is rubbed along the subject's abdomen). 15 minutes will be added to your clinically ordered exams that are completed 4 times a year.

SUMMARY:
To determine if ultrasound measurements can accurately measure the blood pressure of flow across a stent that has been placed in a portal vein to reduce portal vein pressure known as Transjugular Intrahepatic Porto-Systemic shunts or TIPS.

DETAILED DESCRIPTION:
To determine if 3D ultrasound measurements can accurately measure the pressure of blood flow across a stent that has been placed in a portal vein. This has been done in order to reduce portal vein pressure. These shunts are known as Transjugular Intrahepatic Porto-Systemic shunts or TIPS.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female 18 years of age and older
2. Have an existing TIPS (Transjugular intrahepatic porto-systemic shunt)
3. Have an ultrasound ordered by your physician to evaluate your TIPS.
4. Able to read, understand and sign informed consent

Exclusion Criteria:

1. Under 18 years of age
2. Cannot be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-07; Primary Completion 2015-01 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Estimate portal blood flow within a transjugular portosystemic shunt | 4 years
  To determine the number of volumes to achieve a specified variance in the measurement and to determine the reproducibility of the volume flow measurements taken at multiple locations within the stent (3 locations with 3 measurements each for a total of 9 acquisitions).
  The physicians will measure volume flow rate three times at three different locations in the shunt (that being proximal, medial and distal) to determine the reproducibility of the flow estimate.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Novelli, M.D., Principal Investigator — University of Michigan Hospital
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No